CLINICAL TRIAL: NCT03511352
Title: Sedentary Behavior Interrupted: A Randomized Crossover Trial of Acute Effects on Biomarkers of Healthy Aging in the Laboratory (Project 1)
Brief Title: Sedentary Behavior Interrupted: A Trial of Acute Effects on Biomarkers of Healthy Aging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dorothy Sears, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 171547
Record Dates: First submitted 2018-03-26; First posted 2018-04-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Condition (Protocol A) (No Intervention): Following a one-hour sitting run-in period, participants will sit for a 5-hour period including a mid-point bathroom break.
- Frequent Sit-to-Stands (Protocol B) (Experimental): Following a 1-hour sitting run-in period, participants will sit for a 5-hour period including a 2-min stand every 15 min throughout the 5-hr protocol period and a mid-point bathroom break.
  Interventions: Behavioral: Frequent sit-to-stands
- Stand More (Protocol C) (Experimental): Following a 1-hour sitting run-in period, participants will sit for a 5-hour period including 5 8-minute standing breaks, 1 per hour, and a mid-point bathroom break.
  Interventions: Behavioral: Stand More

INTERVENTIONS:
Behavioral: Frequent sit-to-stands — Participants will visit the clinic for a 6-hour monitoring period. Following a 1-hour sitting run-in period, participants will sit for an additional 5-hour period including a 2-min stand every 15 min throughout the 5-hr protocol period. Baseline, mid-point, and end-of-visit bathroom breaks for urine sample collection will be conducted, with additional bathroom breaks allowed as needed.
  Other Names: Protocol B
  Arms: Frequent Sit-to-Stands (Protocol B)
Behavioral: Stand More — Participants will visit the clinic for a 6-hour monitoring period. Following a 1-hour sitting run-in period, participants will sit for an additional 5-hour period including 5 8-minute standing interruptions, 1 per hour. Baseline, mid-point, and end-of-visit bathroom breaks for urine sample collection will be conducted, with additional bathroom breaks allowed as needed.
  Other Names: Protocol C
  Arms: Stand More (Protocol C)

SUMMARY:
This protocol "Sedentary Behavior Interrupted: A randomized crossover trial of acute effects on biomarkers of healthy aging in the laboratory (Project 1)" is part of a National Institutes of Aging Program Grant called "Sedentary Time & Aging Mortality and Physical Function (STAR). The overall purpose of the STAR program to is to better understand how to interrupt sitting time and the consequences for healthy aging in postmenopausal women. This protocol (also referred to Project 1 of the STAR program) is a 3-condition randomized crossover clinical trial of up to 86 postmenopausal women to test whether different interruptions to prolonged sitting improve metabolism.

DETAILED DESCRIPTION:
The specific aims of this protocol include:

Aim 1. To investigate the acute effect of sitting interruption modalities on postprandial glucose and insulin concentrations, compared to prolonged sitting.

Aim 2. To investigate the acute effect of sitting interruption modalities on the physiologic parameters of endothelial function, compared to prolong sitting.

Aim 3. To explore the moderating effect of age.

ELIGIBILITY:
Inclusion Criteria:

* female
* 55 years of age and above
* any ethnicity or race
* screened to sit for 8 or more hours per day, perform less than 60 sit-to-stand transitions per day & engage in less than 20 minutes of moderate-to-vigorous physical activity (MVPA) per day
* BMI 25 - 45 kg/m2
* ambulatory
* medically stable without any health conditions that would inhibit standing or PA;
* able to give informed consent & comply with study protocols;
* able to read, communicate, and write fluently in English;
* able to travel to study visits;
* no menstruation for at least one year;
* not participating or not planning to participate in a physical activity or weight loss program or research study.

Exclusion Criteria:

* Mental state that would preclude complete understanding of the protocol or compliance;
* type 1 diabetes;
* type 2 diabetes using insulin or with poor glycemic control (greater than 10% for all participants);
* poorly controlled hypertension (Systolic Blood Pressure ≥165 or Diastolic Blood Pressure ≥100);
* chronic illness that may be associated with weight change (HIV/AIDS, active cancer, or uncontrolled thyroid disease),
* anemia (hemoglobin ≤11g/dL);
* personal or first-degree relative history of venous thrombosis;
* weight instability in past 3 months (no more than 5% up or down);
* regular use of vasodilator medication and high risk of stroke and/or heart attack (i.e., history of multiple hospitalizations (>2X) in the last 6 months), congestive heart failure, atrial fibrillation, and/or stroke;
* regular use of immunosuppressant or corticosteroid medication;
* blood donation less than 56 days prior to screening visit,
* smoking cigarettes or smoking or ingesting anything, and other use of tobacco products including e-cigarettes.
* diagnosis of orthostatic hypotension

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postprandial glucose | 5 hours
  To investigate the acute effect of sitting interruption modalities on postprandial glucose compared to prolonged sitting.
Insulin | 5 hours
  To investigate the acute effect of sitting interruption modalities on insulin concentrations compared to prolonged sitting.

SECONDARY OUTCOMES:
Flow mediated dilation | 5 hours
  To investigate the acute effect of sitting interruption modalities on flow mediated dilation compared to prolonged sitting
Blood pressure | 5 hours
  To investigate the acute effect of sitting interruption modalities on blood pressure compared to prolonged sitting.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT03511352/ICF_000.pdf